CLINICAL TRIAL: NCT02774096
Title: Cerebral and Spinal Protection of Xenon Post-conditioning in Patients Undergoing Aortic Dissection Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, WeiPing Cheng, Professor；Chief Physician, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WCheng 2014-8-24
Record Dates: First submitted 2016-04-25; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Aortic Dissection
Keywords: Aortic dissection; Cerebral and Spinal Protection; Post-conditioning
MeSH Terms: conditions — Aortic Dissection | interventions — Xenon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group（Ascending aorta） (No Intervention): undergo ascending aorta Dissection Repair and thoracoabdominal aortic Dissection Repair
- Xenon Post-conditioning (Experimental): undergo ascending aorta Dissection Repair and thoracoabdominal aortic Dissection Repair
  Interventions: Drug: xenon

INTERVENTIONS:
Drug: xenon
  Arms: Xenon Post-conditioning

SUMMARY:
With more and more people developing hypertension and atherosclerosis, the morbidity rate of Acute Aortic Dissection（AAD） has been increasing. Emergency surgery is the main treatment for Acute Aortic Dissection. However the secondary injury caused by reperfusion of spinal cord could lead to Catastrophic complications,such as paraplegia, hemiplegia or even death. So spinal protection is always the hot topic in clinical research.

Xenon is an ideal anesthetic gases with the following features,fast onset of action, stable hemodynamics, clean and non-toxic.The animal researches have showed the protective effects of xenon to alleviate the ischemia-reperfusion injury of the nervous system.Those clues suggest that Xenon may have the potential protection of spinal cord in patients undergoing aortic dissection repair.In order to clarify this hypothesis, the investigators designed this randomized, controlled clinic trial to evaluate the protection of Xenon against spinal cord ischemia-reperfusion injury and the potential mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Patients doing selective operation of Bentall and Sun's or partial aortic arch replacement
* Patients doing selective operation of the full chest and abdominal aorta replacement

Exclusion Criteria:

* Emergency patient
* Patients with severe mental and neurological dysfunction
* Patients with severe hearing and visual impairment
* Illiteracy or patients can't cooperate with doing the cognitive function score
* Patients with severe cardiac insufficiency
* critically ill or dying patients
* Patients refuse to sign the informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
mini mental state examination | 18h before the surgery
NIHSS's score | the 1st day after the surgery
ASIA impairment scale（ASIA's score ） | 18h before the surgery
males | 18h before the surgery
age | 18h before the surgery
height | 18h before the surgery
weight | 18h before the surgery
History of Smoking | 18h before the surgery
History of Hypertension | 18h before the surgery
History of Diabetes Mellitus | 18h before the surgery
New York Heart Association Heart function score | 18h before the surgery
duration of cardiopulmonary bypass (CPB) | 1h after the surgery
duration of Aortic cross-clamping | 1h after the surgery
duration of low flow in CPB | 1h after the surgery
duration of stopping the circulation | 1h after the surgery
the lowest nasopharyngeal temperature | 1h after the surgery
the lowest rectal temperature | 1h after the surgery
duration of surgery | 1h after the surgery
duration of recovering of consciousness from the end of the surgery | 3 days after the surgery
duration of extubation from the end of the surgery | 3 days after the surgery
duration in the ICU | 15 days after the surgery
days in hospital | 15 days after leaving hospital
pulmonary infection | 15 days after the surgery
plasma S100β | immediately after anesthesia induction
plasma neuron specific enolase, | immediately after anesthesia induction
plasma myelin basic protein(MBP) | immediately after anesthesia induction
plasma glial fibrillary acidic protein (GFAP) | immediately after anesthesia induction
Cerebrospinal fluid(CSF) S100β | immediately after anesthesia induction
CSF neuron specific enolase(NSE), | immediately after anesthesia induction
CSF MBP | immediately after anesthesia induction
CSF GFAP | immediately after anesthesia induction
CSF Tumor Necrosis Factor-α(TNF-α) | immediately after anesthesia induction
CSF interleukin-10 (IL-10) | immediately after anesthesia induction
CSF IL-6 | immediately after anesthesia induction
CSF IL-2 | immediately after anesthesia induction
somatosensory evoked potential(SEP) | immediately after anesthesia induction
MEP | immediately after anesthesia induction
Mini mental state ex amination | the 7th day after the surgery
NIHSS's score | the 2nd day after the surgery
NIHSS's score | the 3rd day after the surgery
ASIA's score | the 1st day after the surgery
ASIA's score | the 2nd day after the surgery
ASIA's score | the 3rd day after the surgery
plasma S100β | immediately the end of surgery
plasma S100β | the 1st day after the surgery
plasma S100β | the 3rd day after the surgery
plasma S100β | the 7th day after the surgery
plasma neuron specific enolase, | immediately the end of surgery
plasma neuron specific enolase, | the 1st day after the surgery
plasma neuron specific enolase, | the 3rd day after the surgery
plasma neuron specific enolase, | the 7th day after the surgery
plasma MBP | immediately the end of surgery
plasma MBP | the 1st day after the surgery
plasma MBP | the 3rd day after the surgery
plasma MBP | the 7th day after the surgery
plasma GFAP | immediately the end of surgery
plasma GFAP | the 1st day after the surgery
plasma GFAP | the 3rd day after the surgery
plasma GFAP | the 7th day after the surgery
CSF S100β | immediately the end of surgery
CSF S100β | the 1st day after the surgery
CSF S100β | the 2nd day after the surgery
CSF S100β | the 3rd day after the surgery
CSF neuron specific enolase, | immediately the end of surgery
CSF neuron specific enolase, | the 1st day after the surgery
CSF neuron specific enolase, | the 2nd day after the surgery
CSF neuron specific enolase, | the 3rd day after the surgery
CSF MBP | immediately the end of surgery
CSF MBP | the 1st day after the surgery
CSF MBP | the 2nd day after the surgery
CSF MBP | the 3rd day after the surgery
CSF GFAP | immediately the end of surgery
CSF GFAP | the 1st day after the surgery
CSF GFAP | the 2nd day after the surgery
CSF GFAP | the 3rd day after the surgery
CSF TNF-α | immediately the end of surgery
CSF TNF-α | the 1st day after the surgery
CSF TNF-α | the 2nd day after the surgery
CSF TNF-α | the 3rd day after the surgery
CSF IL-10 | immediately the end of surgery
CSF IL-10 | the 1st day after surgery
CSF IL-10 | the 2nd day after surgery
CSF IL-10 | the 3rd day after surgery
CSF IL-6 | immediately the end of surgery
CSF IL-6 | the 1st day after surgery
CSF IL-6 | the 2nd day after surgery
CSF IL-6 | the 3rd day after surgery
CSF IL-2 | immediately the end of surgery
CSF IL-2 | the 1st day after surgery
CSF IL-2 | the 2nd day after surgery
CSF IL-2 | the 3rd day after surgery
SEP | immediately after blocking the aorta
SEP | immediately after opening the aorta
SEP | immediately the end of the surgery
SEP | the 4th hour after back to ICU
MEP | immediately after blocking the aorta
MEP | immediately after opening the aorta
MEP | immediately the end of the surgery
MEP | the 4th hour after back to ICU

CONTACTS AND LOCATIONS:
Overall Officials: WeiPing Cheng, master, Principal Investigator — Chief Physician，Professor

IPD SHARING:
Plan to Share IPD: Undecided